CLINICAL TRIAL: NCT03066700
Title: Prognostic Factors of Outcome in Patient With Malignant Gastrointestinal Bleeding Treated With a Novel Hemostatic Power
Brief Title: Prognostic Factors in Malignant GI Bleeding Treated With Hemostatic Powder
Status: Completed | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Principle investigator, Gastrointestinal Unit, King Chulalongkorn Memorial Hospital
Other Study IDs: RP012
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Death
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemospray application: The patients with GI bleeding from tumor and received Hemospray as a hemostasis method.
  Interventions: Device: Hemostatic powder

INTERVENTIONS:
Device: Hemostatic powder — HemosprayTM (Tc-325) is an endoscopic hemostatis powder that came onto market recently. It is made of an inorganic, non-absorbable powder which acts locally at the mucosa. When spraying the powder on to the bleeding site, it creates an adherent stable barrier sheath that allows for at least temporary hemostasis. Neither luminal nor systemic side effects have been reported to date.
  Other Names: HemosprayTM

SUMMARY:
This is a retrospective study to identify the prognostic factors of the good outcomes in patients who presented with upper GI bleeding from tumor and received Hemospray via endoscopy for hemostatic control. The good outcomes were assessed by immediate hemostasis, rebleeding at 72 hours as well as 7, 14 and 30 days following presentation at initial bleeding episode and also 6-month survival rate.

DETAILED DESCRIPTION:
Tumor-related gastrointestinal (GI) bleeding is increasing due to the advancement of treatment in oncology. However, conventional endoscopic hemostatic methods are not reliable to control bleeding. Surgery, embolization, and radiotherapy can served as the salvage hemostasis; though, a bridging endoscopic therapy is required during resuscitation and stabilization of the patients. Hemospray is a recent novel endoscopic hemostatis powder which has a trend to be an effective instrument for controlling the active upper GI tumor bleeding from a match-pair, case-control study by the author's recent publication. Consequently, the authors hypothesized that there are some prognostic factors related to the outcome of Hemospray treatment in tumor bleeding.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen in the emergency room and/or hospitalized for malignant gastrointestinal haemorrhage from 2011 to 2017

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases will have been treated at the McGill University Health Centre in Montreal, Canada (MUHC; Royal Victoria Hospital - RVH and Montreal General Hospital - MGH sites) and King Chulalongkorn Memorial Hospital (KCMH), Chulalongkorn University, Bangkok, Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 6 months
  Death rate after applying HemosprayTM

SECONDARY OUTCOMES:
Rebleeding rate | 30 days
  Bleeding from tumor after applying HemosprayTM

CONTACTS AND LOCATIONS:
Locations (1):
- King chulalongkorn memorial hospita, Bangkok, Pathum Wan, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pittayanon R, Rerknimitr R, Barkun A. Prognostic factors affecting outcomes in patients with malignant GI bleeding treated with a novel endoscopically delivered hemostatic powder. Gastrointest Endosc. 2018 Apr;87(4):994-1002. doi: 10.1016/j.gie.2017.11.013. Epub 2017 Nov 20. PMID 29158179